CLINICAL TRIAL: NCT01576211
Title: Investigating the Frequency of Loss of Imprinting Across a Birth Cohort and the Link DNA Methylation Plays
Brief Title: Studying Genes Using Cord Blood and Placenta Samples From Relatively Healthy Newborns and Samples From Younger Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B6; COG-AREN12B6 (Other: Children's Oncology Group); CDR0000730596 (Other: Clinical Trials.gov); AREN12B6 (Other: Children's Oncology Group); NCI-2012-00726 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer
Keywords: Wilms tumor and other childhood kidney tumors
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — DNA Methylation; Gene Expression Profiling; Base Sequence; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: allele-specific oligonucleotide real-time quantitative polymerase chain reaction
Genetic: gene expression analysis
Genetic: nucleic acid sequencing
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from newborns and from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies cord blood and placenta tissue from newborns, and tumor tissue samples from patients with Wilms tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* What is the frequency of loss of imprinting at birth (in the cord blood and placenta) in a relatively healthy birth cohort?
* Does deoxyribonucleic acid (DNA) methylation levels at imprinting genes have a direct association to the gene expression?

OUTLINE: Archived tumor tissue, cord blood, and placenta samples are analyzed for DNA methylation, single nucleotide polymorphism, and gene expression by polymerase chain reaction (PCR), pyrosequencing, and quantitative real-time PCR. Information regarding gender and age of the samples are also collected, if possible.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Wilms tumor tissue samples from Caucasians (fresh or frozen), or DNA and ribonucleic acid (RNA) samples already isolated from patients registered on Children's Oncology Group Wilms tumor protocols
* Normal/control blood samples from matched individuals
* Cord blood/ placenta samples from the Michels lab Epigenetic Birth Cohort

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients registered on Children's Oncology Group Wilms tumor protocols
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of loss of imprinting at birth
Association between methylation levels and gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Karin Michels, MD, PhD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center